CLINICAL TRIAL: NCT02715986
Title: Structural-functional Brain Changes in Severely Depressed Patients Before and After Treatment With Electroconvulsive Therapy: an Exploratory Study
Brief Title: Brain Changes in Severely Depressed Patients Before and After Treatment With Electroconvulsive Therapy
Acronym: ECT-IM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/15/7733; 15 7733 02 (Other Grant/Funding Number: University Hospital Toulouse, local funding 2015)
Record Dates: First submitted 2015-12-14; First posted 2016-03-22 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Severe Depression
Keywords: ECT; Diffusion Tensor Imaging (DTI); fMRI
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Severly depressed patients (Experimental): Recruitment of twenty depressive subjects will be conducted within the hospital service adult psychiatry.These patients are referred for indication of ECT sessions for severe resistant depression. Four MRI evaluations (3T MRI examination) are programmed in such patients to analyze structural changes in the hippocampus.
  Interventions: Device: 3T MRI

INTERVENTIONS:
Device: 3T MRI — Four visits will be conducted during the prospective follow during which will be carried out a 3T MRI examination, assessment of assessment of depressive symptomatology and anterograde memory: within 7 days prior to the first session of ECT, within 48 hours after the first ECT session, within 48 hours after the first effective ECT session and within 10 days of the last session of ECT.

SUMMARY:
Electroconvulsive therapy (ECT) is a non-pharmacological treatment used in resistant depression whose effectiveness has been demonstrated. However, the brain mechanisms underlying this therapeutic effect remain unclear. Many animal studies show a neurotrophic action of ECT on the hippocampus: increased neurogenesis, synaptogenesis, proliferation of glial cells. In addition, functional imaging of "resting state" type have shown, among depressed patients after ECT, increased functional connectivity . These results were reinforced by the recent work of Perrin (2012). In view of this a priori contradictory, it seems appropriate to continue research neuroanatomical correlates subtending neurofunctional processes responsible at the same time improving the clinical depressive. The investigators suggest using an original technique never used in this type of population: Functional magnetic resonance imaging (fMRI) or multimodal structural-functional. This method will allow us to study the impact of ECT on brain structures involved in major depressive disorder: hippocampus.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic and Statistical Manual of Mental Disorders-V (DSM) diagnosis of major depressive disorder
* indication of ECT and signing the consent for conducting a ECT
* right-handed
* be of French mother tongue
* belong to a social security scheme
* sign an informed consent

Exclusion Criteria:

* against indication for MRI
* against indication to anesthesia
* processes brain expensive
* pregnant woman
* refuse to be informed of an abnormality detected during MRI
* Patients holders of stimulation electrodes
* presence history of neurological disease
* presence history of head injury
* Mini-Mental State Examination (MMSE) <15/30
* presence of neurodegenerative disease
* patients who have had ECT treatment in the last 6 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Morphological changes in the hippocampus between baseline and after the first ECT effective session as assessed by volume measure in multimodal MRI. | Within 48 hours after the first effective ECT session.
  Visit 3 will take place within 48 hours after the first ECT session effective.

SECONDARY OUTCOMES:
Functional connectivity changes of the hippocampus-related networks between baseline and after the first effective ECT session as assessed by measure of connectivity in multimodal MRI. | Within 48 hours after the first effective ECT session.
  Visit 3 will take place within 48 hours after the first ECT session effective.
Morphological changes of the hippocampus-related networks between baseline and after the first ECT session as assessed by measure of volume in multimodal MRI. | Within 48 hours after the first ECT session.
  Visit 2 will take place within 48 hours after the first ECT session
Morphological changes of the hippocampus-related networks between baseline and after the first ECT session as assessed by average diffusivity in multimodal MRI. | Within 48 hours after the first ECT session.
  Visit 2 will take place within 48 hours after the first ECT session
Functional changes of the hippocampal-related networks between baseline and after the first ECT session as assessed by measure of connectivity in multimodal MRI. | Within 48 hours after the first ECT session.
  Visit 2 will take place within 48 hours after the first ECT session
Morphological changes in the hippocampus and hippocampal-related networks related to ECT between baseline and after remission as assessed by measure of volume in multimodal MRI | Within 10 days after remission.
  Remission is defined by a score of 7 or less on Hamilton Depression Rating
Morphological changes in the hippocampus and hippocampal-related networks related to ECT between baseline and after remission as assessed by | Within 10 days after remission.
  Remission is defined by a score of 7 or less on Hamilton Depression Rating
Functional changes in the hippocampus and hippocampal-related networks related to ECT after remission as assessed by measure of connectivity in multimodal MRI. | Within 10 days after remission
  Remission is defined by a score of 7 or less on Hamilton Depression Rating Scale (HDRS).
Evolution of Real Life/Real Impact-16 (RLRI-16) score after the first ECT, after ECT first "effective" and after remission | Within 7 days before first ECT, after the first ECT, within 48 hours after the first effective ECT and within 10 days after remission
  RLRI-16 test will be realised during all visits, after ECT.
Changes in the intensity of depressive symptoms score (Hamilton Depression Rating Scale) after the first ECT, ECT first "effective" and after remission | Within 7 days before first ECT, after the first ECT, within 48 hours after the first effective ECT and within 10 days after remission
  Hamilton Depression Rating Scale will be realised during all visits, after ECT.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe ARBUS, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Hôpital de psychiatrie, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott CC, Lemke NT, Gopal S, Thoma RJ, Bustillo J, Calhoun VD, Turner JA. Electroconvulsive therapy response in major depressive disorder: a pilot functional network connectivity resting state FMRI investigation. Front Psychiatry. 2013 Mar 1;4:10. doi: 10.3389/fpsyt.2013.00010. eCollection 2013. PMID 23459749
- [Background] Moreaud O, Belliard S, Snowden J, Auriacombe S, Basaglia-Pappas S, Bernard F, Bon L, Boutantin J, Boutoleau-Bretonniere C, Charnallet A, Coutant E, David D, Deramecourt V, Gaestel Y, Garnier S, Guichart E, Hahn-Barma V, Lebail B, Lebrun-Givois C, Lamy E, Le Carret N, Lemesle B, Memin A, Pariente J, Pasquier F, Renou P, Rouaud O, Sarazin M, Thomas-Anterion C, Vercelletto M, Virat-Brassaud ME. [Semantic dementia: reflexions of a French working group for diagnostic criteria and constitution of a patient cohort]. Rev Neurol (Paris). 2008 Apr;164(4):343-53. doi: 10.1016/j.neurol.2008.02.031. Epub 2008 Apr 3. French. PMID 18439926
- [Background] Berman RM, Prudic J, Brakemeier EL, Olfson M, Sackeim HA. Subjective evaluation of the therapeutic and cognitive effects of electroconvulsive therapy. Brain Stimul. 2008 Jan;1(1):16-26. doi: 10.1016/j.brs.2007.08.005. Epub 2007 Dec 3. PMID 20633366
- [Background] Bertolino A, Arciero G, Rubino V, Latorre V, De Candia M, Mazzola V, Blasi G, Caforio G, Hariri A, Kolachana B, Nardini M, Weinberger DR, Scarabino T. Variation of human amygdala response during threatening stimuli as a function of 5'HTTLPR genotype and personality style. Biol Psychiatry. 2005 Jun 15;57(12):1517-25. doi: 10.1016/j.biopsych.2005.02.031. PMID 15953488
- [Background] Blumberg HP, Kaufman J, Martin A, Whiteman R, Zhang JH, Gore JC, Charney DS, Krystal JH, Peterson BS. Amygdala and hippocampal volumes in adolescents and adults with bipolar disorder. Arch Gen Psychiatry. 2003 Dec;60(12):1201-8. doi: 10.1001/archpsyc.60.12.1201. PMID 14662552
- [Result] Yrondi A, Nemmi F, Billoux S, Giron A, Sporer M, Taib S, Salles J, Pierre D, Thalamas C, Schmitt L, Peran P, Arbus C. Significant Decrease in Hippocampus and Amygdala Mean Diffusivity in Treatment-Resistant Depression Patients Who Respond to Electroconvulsive Therapy. Front Psychiatry. 2019 Sep 19;10:694. doi: 10.3389/fpsyt.2019.00694. eCollection 2019. PMID 31607967
- [Result] Yrondi A, Nemmi F, Billoux S, Giron A, Sporer M, Taib S, Salles J, Pierre D, Thalamas C, Rigal E, Danet L, Pariente J, Schmitt L, Arbus C, Peran P. Grey Matter changes in treatment-resistant depression during electroconvulsive therapy. J Affect Disord. 2019 Nov 1;258:42-49. doi: 10.1016/j.jad.2019.07.075. Epub 2019 Jul 31. PMID 31382103